CLINICAL TRIAL: NCT03451864
Title: Maternal 25-hydroxy Vitamin D Level and Adverse Outcomes in Near Term and Full Term Neonates
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Other Study IDs: 29
Record Dates: First submitted 2018-02-25; First posted 2018-03-02 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Neonatal Outcome
MeSH Terms: interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Deficient Vit D: Mothers with serum 25(OH) D levels less than 20 ng/dl
  Interventions: Procedure: Vaginal delivery; Procedure: Cesarean Section
- Normal vit D: Mothers with serum 25(OH) D levels more than 20 ng/dl
  Interventions: Procedure: Vaginal delivery; Procedure: Cesarean Section

INTERVENTIONS:
Procedure: Vaginal delivery — classic vaginal delivery
Procedure: Cesarean Section — routine lower segment cesarean scetion

SUMMARY:
Eighty-eight pregnant women and their newborns were enrolled in a cross-sectional study. Maternal serum 25-OHD was measured by ELISA

DETAILED DESCRIPTION:
Eighty-eight pregnant women and their newborns were enrolled in a cross-sectional study. Maternal serum 25-OHD was measured by ELISA.Maternal 25 (OH) vitamin D measurement: Blood samples for determination of serum 25 (OH) vitamin D were collected by venipuncture and processed as follows: 3 mL blood were collected into plain tubes and allowed to clot for 30 minutes, then it was centrifuged at 1500 round per minute for 15 minutes at room temperature and the serum was separated into clean, properly labeled tubes and stored at ≤ -20°C till assay. Serum 25 (OH) vitamin D level was assessed by Enzyme-Linked ImmunoSorbent Assay (ELISA) using DRG 25-OH Vitamin D (total) ELISA (DRG International, Inc., USA) according to manufacturer's instructions. Vitamin D deficiency is defined by 25(OH) D levels less than 20 ng/d

ELIGIBILITY:
Inclusion Criteria:

* Healthy women Term pregnancy

Exclusion Criteria:

any chronic illness as chronic hypertension or pregestational diabetes pregnancy-related illnesses as preeclampsia, gestational diabetes multiple pregnancy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: 88 full term neonates of both sexes born to 88 healthy women with a mean age was 27.0 ± 5.0 years. Forty-one (46.6%) had normal vaginal delivery and 47 (53.4%) underwent cesarean section
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-24 (Actual)

PRIMARY OUTCOMES:
Neonatal intensive care unit admission | 24 hours after delivery
  Admission of the neonate to NICU

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided